CLINICAL TRIAL: NCT00851227
Title: A Phase 1, Open-Label Study to Assess the Effect of Hepatic Impairment on the Pharmacokinetics of Intravenous Conivaptan
Brief Title: Study to Compare Conivaptan in Subjects With Mild & Moderate Liver Impairment Versus Subjects With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 087-CL-086
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Liver Disease; Hyponatremia
Keywords: Pharmacokinetics; Protein Binding; Conivaptan; Vaprisol; Liver Disease
MeSH Terms: conditions — Liver Diseases; Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Mildly Hepatic Impaired Subjects (Experimental)
  Interventions: Drug: conivaptan hydrochloride
- 2. Moderately Hepatic Impaired Subjects (Experimental)
  Interventions: Drug: conivaptan hydrochloride
- 3. Subjects with Normal Hepatic Function (Experimental)
  Interventions: Drug: conivaptan hydrochloride

INTERVENTIONS:
Drug: conivaptan hydrochloride — intravenous
  Other Names: Vaprisol; YM087

SUMMARY:
A study to compare a 48-hour continuous infusion of conivaptan in subjects with mild and moderate liver impairment versus subjects with normal liver function

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Normal Hepatic Function:

  * Weighs at least 45 kg
  * Body mass index between 18 and 40 kg/m2 inclusive
  * Must have normal hepatic function
* Hepatic Impaired Subjects:

  * Weighs at least 45 kg
  * Meets criteria for mild or moderate hepatic impairment defined by Child-Pugh method
  * Body mass index between 18 and 40 kg/m2 inclusive

Exclusion Criteria:

* Subjects with Normal Hepatic Function:

  * Smokes more than 10 cigarettes per day
  * Known to be HIV positive or has HIV antibodies
  * Has clinically significant history or presence of illness, malignancy, or immunodeficiency
  * Is Hepatitis A, B, or C positive
  * Has had a blood transfusion or donated/lost more than 550ml of blood within 8 weeks of study drug administration
  * History of substance abuse within 6 months prior to screening
* Hepatic Impaired Subjects:

  * Has history or presence of biliary obstruction or biliary disease, hepatic encephalopathy, advanced acidities, portal hypertension, or biliary liver cirrhosis
  * Is hypovolemic or has evidence of orthostatic hypotension
  * Smokes more than 10 cigarettes per day
  * Known to be HIV positive or has HIV antibodies
  * Has clinically significant history or presence of illness, malignancy, or immunodeficiency
  * Has clinically significant history or presence of GI symptoms other than those associated with moderate hepatic impairment
  * Has had a blood transfusion or donated/lost more than 550ml of blood within 8 weeks of study drug administration
  * History of substance abuse within 6 months prior to screening

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Measure PK and protein binding of conivaptan | 5 days

SECONDARY OUTCOMES:
Measure tolerability of conivaptan | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Miami, Florida, United States